CLINICAL TRIAL: NCT03792321
Title: Study on Effects of Testosterone Replacement Therapy in Hypogonadal Type 2
Brief Title: Study on Effects of Testosterone Replacement Therapy in Hypogonadal Type 2 Diabetic Patients" (SETH2)
Acronym: SETH2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Kristina Groti, Principal Investigator; MD, PhD, specialist in Internal medicine, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBCE-KG-2014-1
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Hypogonadism, Male; Diabetes Mellitus, Type 2; Obesity
Keywords: testosterone; hypogonadism; diabetes mellitus; visceral obesity; insulin resistance; metabolic syndrome; NAFLD; endothelial function
MeSH Terms: conditions — Eunuchism; Diabetes Mellitus, Type 2; Obesity; Hypogonadism; Diabetes Mellitus; Obesity, Abdominal; Insulin Resistance; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: 55 patients were divided in two groups. P group patients were receiving placebo throughout the first year of this study and T group patients were receiving testosterone. Both groups were receiving TRT throughout the second year.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Active Comparator): Testosterone arm patients were receiving testosterone undecanoate 1000 mg intramuscular injections two years; according to the protocol every 10 weeks
  Interventions: Drug: Testosterone Undecanoate
- Placebo (Placebo Comparator): Placebo arm patients were receiving placebo throughout the first year of this study and testosterone undecanoate 1000 mg intramuscular injections during second year.
  Interventions: Drug: Testosterone Undecanoate; Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Undecanoate — 1000 mg i.m. every 10 weeks
  Other Names: Nebido
Drug: Placebo
  Arms: Placebo

SUMMARY:
Aim of the study was to investigate the effects of testosterone replacement therapy on components of metabolic syndrome, vascular function and morphology, grade of non-alcoholic fatty liver disease (NAFLD), bone mineral density (BMD) and health-related quality of life.

DETAILED DESCRIPTION:
Studies have shown that approximately 50 % of older obese males, who are being treated for diabetes mellitus type 2, also exhibit low testosterone levels. Hypogonadism negatively affects glycemic control, exacerbates early cardio-vascular disease, causes osteoporosis, erectile disfunction, reduces lean body mass, accelerates the accumulation of visceral fat and leads to obesity.

Patients with diabetes mellitus type 2 and confirmed hypogonadism were enrolled into this randomized, double-blind, placebo-controlled clinical study. Placebo group patients were receiving placebo throughout the first year of this study and Testosterone group patients were receiving testosterone undecanoate during first year. Both groups were receiving testosterone undecanoate throughout the second year of this study.

ELIGIBILITY:
Inclusion Criteria:

* men aged > 35 years
* body mass index > 30 kg/m2
* confirmed hypogonadism
* type 2 diabetes mellitus treated with non-insulin therapy

Exclusion Criteria:

* previously treated hypogonadism
* the 2 diabetes mellitus treated with insulin therapy
* a history of current prostate or breast cancer
* severe benign prostatic hyperplasia
* elevated prostate-specific antigen (PSA > 4.0 lg/l)
* severe heart failure
* acute coronary event or procedure during the six months leading up to the study
* chronic obstructive lung disease
* hypothyroidism
* severe obstructive sleep apnea (OSA)
* active infection
* rheumatoid arthritis

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2015-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Effects of testosterone replacement therapy on glycemic control - fasting plasma glucose (FPG) mmol/l | FPG was measured at baseline, after 12 months and after 24 months
  The primary outcome measure was change in glycemic control - fasting plasma glucose (FPG) mmol/l
Effects of testosterone replacement therapy on glycemic control - glycated hemoglobin A1c (HbA1c) % | HbA1c was measured at baseline, after 12 months and after 24 months
  The primary outcome measure was change in glycemic control - glycated hemoglobin A1c (HbA1c) %
Effects of testosterone replacement therapy on parameters of metabolic syndrome - change in HOMA-IR | HOMA-IR was calculated at the baseline, after 12 months and after 24 months of clinical trial.
  The primary outcome measure was change in Homeostasis model assessment of insulin resistance (HOMA-IR)
Effects of testosterone replacement therapy on vascular function - change in flow mediated dilatation (FMD) % | FMD was measured at baseline, after 12 months and after 24 months
  The primary outcome measure was change in flow mediated dilatation (FMD) % assessed by vascular ultrasound
Effects of testosterone replacement therapy on vascular morphology - intima-media thickness (IMT) | IMT was measured at baseline, after 12 months and after 24 months
  The primary outcome measure was change in intima-media thickness (IMT) mm assessed by vascular ultrasound

SECONDARY OUTCOMES:
Effects of testosterone replacement therapy on non-alcoholic fatty liver disease (NAFLD) | Grade of NAFLD was determined at baseline and after 24 months
  The secondary outcome was change in grade of non-alcoholic fatty liver disease (NAFLD) graded as either "none", "mild", "moderate" and "severe", assessed by abdominal ultrasound
Effects of testosterone replacement therapy on bone mineral density (BMD) | Change in bone mineral density was measured at baseline and after 24 months
  The secondary outcome was change in bone mineral density assessed by dual-energy x-ray absorptiometry (DXA) g/cm^2
Effects of testosterone replacement on total testosterone (TT), calculated free testosterone (cFT), and calculated bioavailable testosterone (BT) concentrations | Changes in total testosterone (TT), calculated free testosterone (cFT), and calculated bioavailable testosterone (BT) concentrations were measured baseline, after 12 months and 24 months
  The secondary outcome were changes in total testosterone (TT), calculated free testosterone (cFT), and calculated bioavailable testosterone (BT) concentrations - all in nmol/l
Effects of testosterone replacement on prostate specific antigen (PSA) | Prostate specific antigen (PSA) was measured at baseline,3,6,12,15,18 and 24 months
  The secondary outcome was change in prostate specific antigen (PSA) ng/ml
Effects of testosterone replacement on hematocrit | Hematocrit was measured at baseline,3,6,12,15,18 and 24 months
  The secondary outcome was change in hematocrit (Hct) %

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Groti Antonic, MD, PhD, Principal Investigator — University Medical Centre Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided